CLINICAL TRIAL: NCT01848756
Title: A Single Arm, Phase 1/2 Study of SNX-5422 in Subjects With Selected HER2 Positive Cancers.
Brief Title: Safety and Efficacy of SNX-5422 in Human Epidermal Growth Factor Receptor 2 (HER2) Positive Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN1-008
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Cancer
Keywords: SNX-5422; HER2 positive cancer
MeSH Terms: conditions — Neoplasms | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SNX-5422 (Experimental): Open-label administration of SNX-5422 capsules to total 100 mg/m2 every other day for 21 days (total = 11 doses), out of a 28-day treatment cycle. Subjects will continue treatment on a 28-day cycle at the discretion of the principal investigator based on safety.
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — Capsule(s) dosed every other day for 21 days (total = 11 doses), out of a 28-day treatment cycle.

SUMMARY:
Hsp90 is a chemical in the body that is involved in the promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90

DETAILED DESCRIPTION:
Heat shock protein 90 (Hsp90) chaperone proteins stabilize well over 200 different known client proteins helping them to fold correctly as they take up their rightful positions in the cell. Hsp90 has a special fondness for oncoproteins whose structures shift according to functional state. Among Hsp90's clients, a surprising number are well recognized targets in oncology, including human epidermal growth factor receptor 2 (HER2). SNX-5422 is a pro-drug of SNX-2112, a potent, highly selective, small-molecule inhibitor of the molecular chaperone heat shock protein 90 (Hsp90). Treatment of HER2-positive cell lines such as BT-474 with the Hsp90 inhibitor SNX-2112 results in cellular degradation, decreased levels of phospho-AKT/cyclin D1, and increased apoptosis. Furthermore, treatment with SNX-5542 caused tumor regression, including remission in a HER2-overexpressing breast cancer xenograft model. SNX-5422 has demonstrated significant antitumor activity in mouse xenograft models of various human malignancies, including breast (BT474, MX-1), lung (H1975, H1650, EBC-1), colon (HT29), prostate (PC3), and melanoma (A375) with multiple oral dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females .
* Confirmed diagnosis of locally advanced or metastatic breast, esophagogastric, urothelial, or non-small cell lung cancer.
* Histological or cytological confirmed carcinoma with HER2 amplification (IHC 3+ or FISH+ (>2 HER2:CEP17)).
* Subjects with advanced or metastatic breast cancer must have received no more than 5 prior lines of anticancer therapy, including trastuzumab (but excluding hormonal treatments).
* Subjects with advanced or metastatic HER2 positive esophagogastric cancer must have received no more than 5 prior lines of anticancer therapy, including trastuzumab.
* Subjects with advanced or metastatic, urothelial carcinoma or non-small cell lung cancer must have received at least one, but no more than 5 prior lines of anticancer therapy.
* Measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Life expectancy of at least 3 months.
* Karnofsky performance score ≥70.
* Adequate baseline laboratory assessments
* Recovered from toxicities of previous anticancer therapy, with the exception of CTCAE grade 1 sensory neuropathy.

Exclusion Criteria:

* Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable
* Prior treatment with any Hsp90 inhibitor.
* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable disease.
* Major surgery within 4 weeks prior to first dose of SNX-5422.
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation).
* The need for treatment with medications with clinically-relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422.
* Screening ECG QTc interval ≥470 msec for females, ≥450 msec for males.
* At increased risk for developing prolonged QT interval
* Patients with chronic diarrhea or with grade 2 or greater diarrhea despite maximal medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption, including gastric bypass.
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* Known seropositive for human immunodeficiency virus (HIV) or hepatitis C virus (HCV).
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Treatment with other anticancer drugs within 28 days or 5 half-lives of anticancer therapy (whichever is shorter), and treatment with any other investigational agent is prohibited from 30 days prior to the first dose of SNX-5422 and throughout the study
* Glaucoma, retinitis pigmentosa, macular degeneration, or any retinal changes detected by ophthalmological examination.
* Other serious concurrent illness or medical condition.
* Psychological, social, familial, or geographical reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNX-5422
Started | 15
Completed | 12 (Cycle 1)
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Enrolled in Error | 1

BASELINE CHARACTERISTICS:
Arm/Group | SNX-5422
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.9)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The effect of SNX-5422 on tumor progression. Objective tumor responses (complete remissions plus partial remissions) and clinical benefit rate (complete remissions plus partial remissions plus stable disease at 6 months) will be listed by subject. Tumor measurements made using Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Up to 24 months from last patient entry
Population: Per protocol population including all enrolled evaluable subjects.Due to slow recruitment and availability newer targeted treatments the study was terminated for business reasons. No patient completed 6 months on study, the first analysis time point for this endpoint, at the time of study termination
Arm/Group | SNX-5422
Number analyzed (Participants) | 0

2. Primary Outcome: Progression Free Survival
Description: Time on treatment with at worst stable disease.
Time Frame: Every 3 months until 24 months after the last subject has been enrolled
Population: Due to slow recruitment and availability newer targeted treatments the study was terminated for business reasons. No patient completed 3 months on study, the first analysis time point for this endpoint, at the time of study termination
Arm/Group | SNX-5422
Number analyzed (Participants) | 0

3. Primary Outcome: Overall Survival
Description: Time from start of treatment that patients remain alive.
Time Frame: Every 3 months until 24 months after the last subject has been enrolled
Population: as for outcome 2
Arm/Group | SNX-5422
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of patients experiencing treatment emergent adverse events.
Time Frame: Day 28 of each cycle
Population: All Treated Subjects
Measure: Number; unit: participants
Arm/Group | SNX-5422
Number analyzed (Participants) | 15
participants | 15

5. Secondary Outcome: Changes in Vital Signs, Physical Examination or Clinical Laboratory From Baseline
Description: Descriptive summaries of vital signs, physical examination and clinical laboratory changes will be presented by treatment received.
Time Frame: Day 28 of each cycle
Population: All Treated Subjects
Measure: Number; unit: participants
Arm/Group | SNX-5422
Number analyzed (Participants) | 15
participants
  All laboratory abnormalities | 8
  ALT/AST increases | 6
  Alkaline phosphatase increase | 3
  Vital signs | 0
  Systolic/diastolic blood pressure | 0
  Respiratory rate | 0
  Temperature | 0
  ECG | 0

6. Secondary Outcome: Ophthalmologic Changes From Baseline
Description: Ophthalmologic assessments will be presented by cohort, study visit and dose. Number of subjects experiencing clinically relevant changes from baseline in any of these examinations will be presented using descriptive summary
Time Frame: Screening, end of Cycle 1, final visit
Population: ll Treated Subjects
Measure: Number; unit: participants
Arm/Group | SNX-5422
Number analyzed (Participants) | 15
participants | 1

7. Secondary Outcome: Adverse Events by Severity and Relationship to Treatment
Description: Number of patients experiencing adverse events by highest recorded severity and relationship to study tretament
Time Frame: Every 28 day cycle
Population: All treated subjects
Measure: Number; unit: participants
Arm/Group | SNX-5422
Number analyzed (Participants) | 15
participants
  Subjects with adverse events | 15
  Subjects with Grade 3 or 4 adverse events | 8
  Subjects with Grade 5 adverse events | 2
  Subjects with treatment related adverse events | 15
  Subjects with Grade 3 or 4 AEs related to treatmen | 7
  Subjects with Grade 5 AEs related to treatment | 0

ADVERSE EVENTS:
Time Frame: From patient screening to removal from study, average time on study 49+/-16 days
Description: Regular Investigator Assessment including patient volunteered reports
Arm/Group | SNX-5422
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SNX-5422 (N=15)
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cardiac Tamponade (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Asthenia (General disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SNX-5422 (N=15)
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
hyponatraemia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 6
Chills (General disorders) | 1
Mucosal Inflammation (General disorders) | 1
Aspartate Aminotransferase increased (Investigations) | 5
Alanine Aminotransferase Increased (Investigations) | 3
Blood Alkaline Phosphatase Increased (Investigations) | 2
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Blood Cholesterol Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Vision Blurred (Eye disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less